CLINICAL TRIAL: NCT06642155
Title: Testing the Efficacy of ResponsiblePlay©: MTM-Based Intervention for Responsible Gambling for College Students
Brief Title: Theory-based Intervention for Promoting Responsible Gambling Among College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Manoj Sharma, Professor & Chair, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNLV-2024-507
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Problem Gambling; Pathological Gambling; Behavioral Addiction; Gambling Disorder
Keywords: Responsible Gambling; College Students; Problem Gambling; Pathological Gambling; Behavioral Interventions; Health Behavior Change; Multi-theory Model (MTM); Randomized Controlled Trial (RCT); Public Health Intervention; Gambling Disorder Prevention
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups-the MTM-based ResponsiblePlay© intervention group and the knowledge-based intervention group, which will run in parallel.
Who Masked: Participant
Masking Description: The participants will not be aware of whether they are receiving the ResponsiblePlay© intervention or the knowledge-based intervention. This single-blind design helps reduce bias related to participants' expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RESPONSIBLEPLAY© MTM-Based Intervention (Experimental): Participants will receive a theory-based intervention designed to promote responsible gambling behaviors using the Multi-theory Model (MTM) of health behavior change. The intervention focuses on both the initiation and sustenance of responsible gambling through six constructs:
  Participatory Dialogue: Discussing the pros and cons of responsible gambling. Behavioral Confidence: Building confidence to practice responsible gambling. Changes in the Physical Environment: Modifying surroundings to limit gambling opportunities.
  Emotional Transformation: Managing emotions to maintain behavior change. Practice for Change: Planning and practicing responsible gambling strategies. Changes in the Social Environment: Leveraging support from family, friends, and professionals.
  This intervention aims to provide practical strategies for adopting and maintaining responsible gambling behaviors.
  Interventions: Behavioral: RESPONSIBLEPLAY© MTM-Based Intervention
- Knowledge-Based Intervention (Active Comparator): Participants will receive educational content about the risks of gambling and strategies for responsible gambling in the form of lectures and reading materials.
  Interventions: Behavioral: Knowledge-Based Intervention

INTERVENTIONS:
Behavioral: RESPONSIBLEPLAY© MTM-Based Intervention — Participants in this group will receive a theory-based intervention using the Multi-theory Model (MTM) of health behavior change. The intervention includes participatory dialogue, behavioral confidence-building, and strategies to modify the physical and social environments. It also incorporates emotional transformation and practice for change. Sessions will be delivered in-person over three weeks, focusing on promoting responsible gambling behaviors.
  Arms: RESPONSIBLEPLAY© MTM-Based Intervention
Behavioral: Knowledge-Based Intervention — Participants in this group will receive a knowledge-based intervention that provides information on gambling risks and responsible gambling strategies. The intervention consists of lectures and reading materials delivered in-person over three weeks. It focuses on raising awareness of gambling risks but does not include the behavioral change strategies used in the MTM-based intervention.
  Arms: Knowledge-Based Intervention

SUMMARY:
The goal of this clinical trial is to learn if the RESPONSIBLEPLAY© intervention helps promote responsible gambling behaviors in University of Nevada, Las Vegas (UNLV) students aged 21 and older who have a Problem Gambling Severity Index (PGSI) score of 3 or higher. The main questions it aims to answer are:

Does the intervention reduce harmful gambling behaviors? Does the intervention increase responsible gambling practices? Researchers will compare participants receiving the RESPONSIBLEPLAY© intervention with those receiving a knowledge-based intervention to see if the RESPONSIBLEPLAY© intervention is more effective.

Participants will:

Attend three face-to-face sessions on responsible gambling over three weeks. Complete surveys before, after, and eight weeks after the intervention to track their progress.

DETAILED DESCRIPTION:
This study investigates the efficacy of the RESPONSIBLEPLAY© intervention, designed to promote responsible gambling behaviors among college students at UNLV. College students are a vulnerable group for developing gambling-related problems, with a significantly higher prevalence of problem and pathological gambling compared to the general population. This randomized controlled trial (RCT) will compare the RESPONSIBLEPLAY© intervention, which is based on the Multi-theory Model (MTM) of health behavior change, to a traditional knowledge-based intervention.

The RESPONSIBLEPLAY© intervention addresses both the initiation and sustenance of behavior change, incorporating elements such as participatory dialogue, behavioral confidence, and changes in the social and physical environments. The intervention aims to equip participants with practical strategies to manage and limit gambling behaviors.

The study will take place over a three-week period, with face-to-face sessions designed to engage participants in discussions and self-guided activities that promote responsible gambling. Follow-up assessments will be conducted at eight weeks post-intervention to evaluate the long-term impact of the intervention. A two-factor repeated measures analysis will be used to assess changes in gambling behaviors and related psychological constructs over time.

The findings from this study may provide critical evidence to support the use of theory-based interventions to reduce gambling-related harms in a college student population, which can inform future public health strategies.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 21 years old.
* Must be a enrolled UNLV student.
* Must engage in gambling activities.
* Must have a score of 3 or higher on the Problem Gambling Severity Index (PGSI), indicating at-risk or problem gambling behavior.

Exclusion Criteria:

* Participants currently receiving treatment for gambling disorders.
* Individuals with cognitive impairments that would affect their ability to provide consent or participate in the intervention.
* Individuals who are not fluent in English (since the intervention materials and assessments will be conducted in English).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in Problem Gambling Severity Index (PGSI) Score | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  The primary outcome will assess changes in the Problem Gambling Severity Index (PGSI) scores, which measure the severity of gambling behavior. The PGSI includes 9 items with a score range of 0 to 27, where higher scores indicate more severe gambling issues. Scores will be collected at baseline, immediately post-intervention, and at an eight-week follow-up.

SECONDARY OUTCOMES:
Change in Participatory Dialogue (Perceived Advantages Minus Perceived Disadvantages) for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in the Participatory Dialogue construct by assessing both perceived advantages and perceived disadvantages of responsible gambling.
  Perceived Advantages will be measured using 5 items (questions 12-16) scored from 0 (not at all likely) to 4 (completely likely), with a possible score range of 0 to 20.
  Perceived Disadvantages will be measured using 5 items (questions 17-21) scored from 0 (not at all likely) to 4 (completely likely), with a possible score range of 0 to 20.
  The overall Participatory Dialogue score is calculated by subtracting the perceived disadvantages score from the perceived advantages score, yielding a possible range from -20 to +20.
Change in Behavioral Confidence for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in Behavioral Confidence using 4 items (questions 22-25) that assess participants' confidence in engaging in responsible gambling. Items are scored on a 5-point Likert scale from 0 (not at all confident) to 4 (completely confident), with a possible total score ranging from 0 to 16 units.
Change in the Physical Environment for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in Changes in the Physical Environment using 3 items (questions 26-28) that assess participants' ability to avoid gambling environments and resist access to gambling resources. Items are scored on a 5-point Likert scale from 0 (not at all sure) to 4 (completely sure), with a possible total score ranging from 0 to 12 units.
Change in Emotional Transformation for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in Emotional Transformation using 3 items (questions 29-31) that assess participants' ability to manage their emotions and stay motivated toward responsible gambling. Items are scored on a 5-point Likert scale from 0 (not at all sure) to 4 (completely sure), with a possible total score ranging from 0 to 12 units.
Change in Practice for Change for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in Practice for Change using 3 items (questions 32-34) that assess participants' ability to maintain responsible gambling behaviors. Items are scored on a 5-point Likert scale from 0 (not at all sure) to 4 (completely sure), with a possible total score ranging from 0 to 12 units.
Change in the Social Environment for Responsible Gambling | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure changes in Changes in the Social Environment using 3 items (questions 35-37) that assess participants' ability to seek support from their social network. Items are scored on a 5-point Likert scale from 0 (not at all sure) to 4 (completely sure), with a possible total score ranging from 0 to 12 units.
Change in Initiation of Responsible Gambling Behaviors | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure the overall Initiation using 3 items (questions 38-40) assessing participants' likelihood of initiating responsible gambling. Items are scored on a 5-point Likert scale from 0 (not at all likely) to 4 (completely likely), with a possible total score range of 0 to 12 units.
Change in Sustenance of Responsible Gambling Behaviors | Baseline, immediately post-intervention (Week 3), and eight-week follow-up (Week 11)
  This outcome will measure the overall Sustenance using 3 items (questions 41-43) assessing participants' likelihood of continuing responsible gambling. Items are scored on a 5-point Likert scale from 0 (not at all likely) to 4 (completely likely), with a possible total score range of 0 to 12 units.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sharma, PhD, Principal Investigator — University of Nevada, Las Vegas (UNLV)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) that underlie the results reported in published articles will be shared, including data dictionaries. Data will be anonymized to protect participant privacy.